CLINICAL TRIAL: NCT02038868
Title: Double-Blind, Placebo-Controlled, Active-Referenced, Parallel-Group Comparative Study in Patients With Benign Prostatic Hyperplasia
Brief Title: A Study to Evaluate the Efficacy and Safety of ASP4901 in Patients With Benign Prostate Hyperplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4901-CL-0201
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Benign Prostate Hyperplasia
Keywords: ASP4901; BPH
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ASP4901 group (Experimental): After the main enrollment, patients will receive an oral dose of ASP4901 once daily for 4 weeks (double-blind treatment period).
  Interventions: Drug: ASP4901
- Placebo group (Placebo Comparator): After the main enrollment, patients will receive an oral dose of placebo once daily for 4 weeks (double-blind treatment period).
  Interventions: Drug: Placebo
- Tamsulosin group (Active Comparator): After the main enrollment, patients will receive an oral dose of tamsulosin once daily for 4 weeks (double-blind treatment period).
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: ASP4901 — oral
  Arms: ASP4901 group
Drug: Tamsulosin — oral
  Other Names: YM617; Harnal
  Arms: Tamsulosin group
Drug: Placebo — oral
  Arms: Placebo group

SUMMARY:
The purpose of this study is to compare the efficacy of ASP4901 with placebo in patients with benign prostatic hyperplasia. The safety and tolerability of ASP4901 will also be evaluated.

DETAILED DESCRIPTION:
This is a multicenter, randomized, parallel-group, placebo-controlled, active-referenced, double-blind study. After obtaining the written consent, patients meeting the eligibility criteria at the preliminary enrollment will receive oral administration of placebo in a single-blinded manner (single-blind placebo run-in period). Then, patients meeting the eligibility criteria at the main enrollment will receive drug or placebo (double-blind treatment period) for 4 weeks. Furthermore, patients will be followed up for 1 week to confirm the safety of the study drugs after the treatment period (safety follow-up period).

ELIGIBILITY:
Inclusion Criteria:

* dysuria associated with BPH for at least 12 weeks before providing consent
* a total IPSS core of 13 or higher
* a QOL score of 3 or higher
* a maximum urinary flow rate (Qmax) of ≥4 mL/sec and <15 mL/sec.
* a prostate volume of ≥20 mL.

Exclusion Criteria:

* A postvoid residual volume (PVR) of >350 mL
* A previous or concurrent symptomatic urinary tract infection within 4 weeks of the study
* A cataract operation scheduled to be performed during the study period
* Previous or concurrent clinically relevant cardiovascular or cerebrovascular disorder within 24 weeks prior to the study
* Hypersensitivity to ASP4901 or tamsulosin hydrochloride
* Presence of serious hepatic diseases, renal diseases, immunological diseases, or pulmonary diseases that are clinically relevant

Ages: 40 Years to 74 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2013-07-22 (Actual); Primary Completion 2014-04-04 (Actual); Study Completion 2014-04-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in total IPSS (International Prostate Symptom Score) | baseline and at the final evaluation (up to 5 weeks)

SECONDARY OUTCOMES:
Change from baseline in each symptom score of IPSS | baseline and at the final evaluation (up to 5 weeks)
Change from baseline in IPSS QOL (quality of life) score | baseline and at the final evaluation (up to 5 weeks)
Proportion of IPSS responder | baseline and at the final evaluation (up to 5 weeks)
  "IPSS responder" is defined as 25% improvement in IPSS
Plasma concentration of ASP4901 | up to 5 weeks
  only for ASP4901 group
Safety assessed by the incidence of adverse events, vital signs, labo-tests and 12-lead ECGs | up to 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (2):
- Japan (2):
  - Kansai
  - Kanto

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=291